CLINICAL TRIAL: NCT06260059
Title: Efficacy of Sodium Glucose Transporter Inhibitor (SGLT2i) in Adult Patients With Congenital Heart Disease
Acronym: EmpaCHD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Anita Saraf (Other)
Collaborators: The Pittsburgh Foundation (Other)
Responsible Party: Sponsor-Investigator, Anita Saraf, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY23070148; Pitt2024 (Other Grant/Funding Number: Pittsburgh Foundation)
Record Dates: First submitted 2024-01-02; First posted 2024-02-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Adult Congenital Heart Disease; Heart Failure
Keywords: congenital heart disease; reduced exercise capacity; decreased cardiac function
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Group 1: Empagliflozin 10 MG daily Group 2: Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin 10 MG (Experimental): Empagliflozin 10 mg daily will be administered for 1 year. The patient and the PI will be blinded (unaware) of the group they are assigned to.
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): Placebo for 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Patient will be given 10 mg of Empagliflozin if randomized to the drug arm or will receive placebo drug for 1 year
  Other Names: Jardiance, Empagliflozin
  Arms: Empagliflozin 10 MG
Drug: Placebo — To patients randomized to the placebo group, a placebo pill will be given
  Other Names: Placebo Drug
  Arms: Placebo

SUMMARY:
The goal of the study is to investigate the feasibility and benefit of novel guideline-directed heart failure therapy drug Empagliflozin (Jardiance) for adult patients with congenital heart disease (ACHD).

DETAILED DESCRIPTION:
As CHD adolescents transition to adulthood, it is becoming evident that in addition to their structural cardiac abnormalities, they also have an intrinsic disease of the heart muscle which manifests as abnormal heart rhythm (arrhythmia) and decreased function (heart failure).

The lifesaving cardiac surgeries during childhood can also contribute to this dysfunction (cardiomyopathy). Hence, patients with CHD require multiple interventions and close clinical follow-up throughout their life. Currently, there are over 2.5 million CHD patients in the U.S. alone, and an additional 40,000 babies are born with CHD every year. Up to 50% of these patients require inpatient hospital care at some point due to their cardiomyopathy.

High-risk ACHD patients do not receive treatment until they present with heart failure or arrhythmia, at which time there is significant evidence of myocardial disease and dysfunction.

Empagliflozin (Jardiance) is an FDA-approved drug that significantly reduces hospitalization risk and cardiovascular death in adult patients with non-CHD heart failure. Studies show that Empagliflozin protects the heart from inflammation, and preliminary evaluation of Empagliflozin in symptomatic ACHD patients showed improved cardiac function and a reduction in heart failure including decreased shortness of breath and increased functional capacity. Empagliflozin as a preventative therapy may delay the onset of comorbidities by reducing inflammation in ACHD patients.

The study hypothesis is that the administration of once-a-day oral Jardiance (Empagliflozin) medication for one year reduces arrhythmia and cardiomyopathy and lowers serum circulating inflammatory factors and improves neurocognitive outcomes in susceptible ACHD patients.

1. Does Empagliflozin 10 milligrams (MG) improve cardiac function in ACHD patients
2. Does Empagliflozin 10 milligrams (MG) improve functional status in ACHD patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of Congenital Heart Disease
* Age 18+
* ACHD level of structural complexity II or III
* Recent (<6 months) decrease in systemic Ejection Fraction (confirmed by cardiac Echocardiogram, Computed Tomography or cMRI) to EF < 60%
* Recent decrease in systemic ejection fraction confirmed by cardiac Echo, CT or MRI by > 5% in the last 6 months or less.
* Must be able to complete neurocognitive assessments on a handheld computer.

Exclusion Criteria:

* Diagnosed with Diabetes
* Contraindication to Jardiance/Entresto or any heart failure medication (per guideline-directed therapy, 2022).
* Previous therapy with Jardiance at <4 weeks
* Glomerular Filtration Rate <20
* Pregnancy, breastfeeding, or planning to become pregnant in the coming year
* History of liver disease - including non-alcoholic fatty liver disease (NAFLD) and cirrhosis
* History of inborn error(s) of metabolism (including but is not exclusive of Glycogen storage disease type 1)
* Glucose-galactose malabsorption, familial hyperinsulinism, maple syrup urine disease,
* Gaucher disease,
* Tay-Sachs disease,
* Mucolipidosis IV,
* Niemann-Pick disease,
* Type A mitochondrial disease,
* Metabolic disorders related to glucose metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Ejection fraction (EF) | Change from baseline in ejection fraction at 1-year
  Cardiac Magnetic Resonance Imaging (cMRI) and echocardiography will be used to measure ventricular function
Change in Myocardial characteristics (T1 mapping of cMRI) | Change from baseline in T1 mapping at 1-year
  Cardiac Magnetic Resonance Imaging (cMRI) without contrast will be used to measure myocardial characteristics
Change in Myocardial characteristics (Global strain on MRI) | Change from baseline of global strain on MRI at 1 year
  Cardiac Magnetic Resonance Imaging (cMRI) will be used to measure myocardial characteristics
Change in Myocardial characteristics (Global strain on echocardiogram) | Change from baseline of global strain on echocardiogram at 1 year
  Echocardiography will be used to measure myocardial characteristics such as global longitudinal strain
Change in functional exercise capacity of participants. | Change from baseline of exercise capacity at 1-year
  Cardiopulmonary exercise stress testing (CPET) will be used to measure functional change in MVO2, RER, Exercise time, METs, and vitals.
Number of Participants Hospitalized for Cardiac Reasons or heart transplantation | Cardiac hospitalizations or transplantation at 1 year.
  Hospitalization for cardiac reasons or heart transplantation
Number of Deaths | Number of deaths at 1 year
  Number of patients who died during the study from all causes

SECONDARY OUTCOMES:
Change in inflammatory serum biomarkers | Change from baseline of serum biomarkers at 1-year
  Serum inflammatory markers will be measured using ELISA assays (R&D systems) to test for change in inflammatory response. Biomarkers tested include IL6, TNF-alpha, GDF-15, and IL10. All biomarkers will be measured in pg/mL. All The biomarkers will be used predictively with clinical changes to assess correlation.
Change in functional Neuropsychological Testing | Change from baseline of neuropsychological testing at 1-year
  NIH toolbox Cognitive battery (for ages 7-85) will be used to evaluate change in neuropsychological function. These tests include:
  Picture Vocabulary Test Oral Reading Recognition List Sorting Working Memory Test Pattern Comparison Processing Speed Test Picture Sequence Memory Test Flanker Inhibitory Control and Attention Test Dimensional Change Card Sort Test
  The Cognition Battery produces three composite scores. A score of 100 is average
  1. Fluid Cognition Composite Score: A global assessment of individual and group fluid cognition functioning.
  2. Crystallized Cognition Composite Score: A global assessment of individual and group verbal cognition.
  3. Cognitive Function Composite Score: It provides a snapshot of general cognitive 15 functioning.
  (the above description of tests is directly extracted from https://www.nihtoolbox.org)
Change in New York Heart Association (NYHA) Class | Change from baseline of NYHA Class at 1-year.
  Subjective perception of functional capacity with NYHA Class I patients reporting no symptoms with exercise and rest to NYHA Class IV patients reporting symptoms at rest.
Change Patient-Reported Outcomes Measurement Information System (PROMIS) | Change from baseline of PROMIS composite score at 1 year
  PROMIS measures patient-reported outcomes (PROs), such as pain, fatigue, physical functioning, emotional distress, and social role participation that have a major impact on quality-of-life across a variety of chronic diseases. PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment, Scores 2.0 SD or more worse than the mean = severe symptoms/impairment
  (information directly extracted from https://sphsoutcomes.net/promis-scoring)
Change in Kansas City Cardiomyopathy (KCCQ) | Change from baseline of KCCQ score at 1 year
  The responses are categorized under 3 subscales (symptom burden, physical limitation and quality of life) with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The total KCCQ score represents the mean of the three subscale scores.
  (Extracted from https://www.ncbi.nlm.nih.gov)
Change in Neuro-QOL | Change from baseline of Neuro-QOL score at 1 year
  Neuro-QoL measures quantify the physical, mental, and social effects experienced by adults and children living with neurological conditions. Function scales, the range of responses is 0 to 4, with 0 being the worst possible total score and 80 being the best.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Saraf, MD, PhD, Principal Investigator — Assistant Professor
Locations (3):
- United States (3):
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Plan to not share individual participant data